CLINICAL TRIAL: NCT02006550
Title: Interrogation of Wnt, Notch and Hedgehog Activity in Primary Tumor Samples
Status: Terminated | Type: Observational
Why Stopped: Lack of Resources and Personnel
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Anthony Capobianco, Professor, University of Miami
Other Study IDs: 20100200
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Cancer
Keywords: Wnt; Notch; Hedgehog; Tumor Sample
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer results when undifferentiated cells grow in an uncontrolled manner, crowding out normal cells, causing morbidity and ultimately mortality. The cancer stem cell theory suggests that most tumors undergo a process of differentiation through which a relatively rare cancer stem or progenitor cell (CSC) gives rise to more differentiated populations of cells (including transiently amplifying cells) comprising the bulk of the tumor. As a result of this cellular diversity, one or more cells within the tumor are likely to be resistant to therapy. Among cells resistant to a given therapy, only CSCs can repopulate the tumor. A key feature of this resistant subset of CSCs is that they repopulate a tumor resistant to the original intervention. The cellular programs driving the uncontrolled proliferation of many solid tumors result from aberrant activity of Wnt, Shh, and/or Notch signaling pathways in CSC. Thus, therapies that down-regulate the activity of these fundamental pathways in CSCs will be effective in the treatment of cancer. The investigators' research program focuses on the elucidation of signaling mechanisms, control of cellular processes and discovery of small molecules that selectively target Wnt, Shh, and Notch signaling pathways that are fundamental to CSCs. Our preliminary results identified a novel Notch associated protein NACK that functions as a transcriptional co-activator of Notch. Moreover, Nack is expressed in human solid tumors and is required for cell survival and tumor growth in notch -dependent tumor cells. The investigators' aim is to further interrogate the link between Notch and Nack.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a primary cancer tumor scheduled for a surgery to remove it.

Exclusion Criteria:

* Patients not diagnosed with a primary cancer scheduled for a standard of care (SOC) surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These are samples derived from discarded tissue obtained through the routine surgical resection of tumors
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2010-06-16 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Identify and isolate the cancer stem cell populations from primary tumor samples. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Capobianco, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States